CLINICAL TRIAL: NCT01104025
Title: An Open Label Phase II Pilot Study of Hybrid ImmunoTherapy(ATG/Dexamethasone/Etoposide) for Hemophagocytic LymphoHistiocytosis:HIT-HLH
Brief Title: Hybrid Immunotherapy for Hemophagocytic LymphoHistiocytosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIT-HLH
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Hemophagocytic Lymphohistiocytosis
Keywords: hemophagocytic lymphohistiocytosis; hybrid immunotherapy; dexamethasone; Etoposide; ATG,rabbit
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — thymoglobulin; Etoposide; etoposide phosphate; Methotrexate; Hydrocortisone; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Induction Therapy (Experimental): ATG, rabbit: intravenous, 5 mg/kg/dose, 5 consecutive days Dexamethasone: intravenous, 20mg/m2/day x7days, 10mg/m2/day x7days, 5mg/m2/day x14days, 2.5mg/m2/day x14days, 1.25mg/m2/day x14days Etoposide: intravenous, 150 mg/m2 weekly, starting 7 days after first dose of Thymoglobulin Methotrexate and hydrocortisone: intrathecal to patients with central nervous system involvement, age< 1 yr: 6/8mg (MTX/HC), 1-2 yrs: 8/10mg, 2-3 yrs: 10/12mg, >3 yrs: 12/15 mg, on day 7, 14, 21 and 42
  Interventions: Drug: ATG, rabbit; Drug: Etoposide; Drug: Methotrexate; Drug: hydrocortisone; Drug: Dexamethasone

INTERVENTIONS:
Drug: ATG, rabbit — ATG, rabbit (Thymoglobulin, Genzyme) will be dosed at 5 mg/kg/dose, given IV on 5 consecutive days (titrated over 4 to 8 hours).
  Other Names: Thymoglobulin
Drug: Etoposide — Etoposide will be dosed at 150mg/m2, given IV. The first dose will be given 7 days (+/- 2 days) after the first dose of ATG, and be given weekly for a total of 7 doses.
  Other Names: Etopophos; Toposar; VePesid
Drug: Methotrexate — Intrathecal Methotrexate and hydrocortisone will be administered to CNS+ patients (CNS+ patients are those patients which have any of the following: elevated CSF (cerebral spinal fluid) protein or white count, seizures, focal or global neurologic deficit, MRI abnormalities consistent with CNS involvement by HLH.) in the following doses: age< 1 yr: 6/8mg (MTX/HC), 1-2 yrs: 8/10mg, 2-3 yrs: 10/12mg, >3 yrs: 12/15 mg. It will be administered (+/- 3 days) on day 7, 14, 21 and 42.
Drug: hydrocortisone — Intrathecal Methotrexate and hydrocortisone will be administered to CNS+ patients (CNS+ patients are those patients which have any of the following: elevated CSF (cerebral spinal fluid) protein or white count, seizures, focal or global neurologic deficit, MRI abnormalities consistent with CNS involvement by HLH.) in the following doses: age< 1 yr: 6/8mg (MTX/HC), 1-2 yrs: 8/10mg, 2-3 yrs: 10/12mg, >3 yrs: 12/15 mg. It will be administered (+/- 3 days) on day 7, 14, 21 and 42.
Drug: Dexamethasone — will be started with the ATG. It will be divided BID, given IV for at least 1 week before switching to PO. Dosing: 20mg/m2/day x7days, 10mg/m2/day x7days, 5mg/m2/day x14days, 2.5mg/m2/day x14days, 1.25mg/m2/day x14days.

SUMMARY:
Despite good progress during the last decade, hemophagocytic lymphohistiocytosis (HLH) remains difficult to treat. Two different treatment regimens have been used successfully. The first one, a treatment regimen based on two drugs called etoposide and dexamethasone, has been used worldwide. The second regimen, based on two drugs called Anti-thymocyte globulin (ATG) and prednisone, has been used mostly at one hospital in Paris, for over 15 years. With either regimen, about three quarters of treated children survive the most difficult time, the first two months after diagnosis. These two different regimens appear to work somewhat differently, and we suspect that combining them may give better results than either regimen alone. We are conducting this clinical trial to test the combination of ATG, dexamethasone, and etoposide for the treatment of HLH.

The purpose of this research study is to find out what effects (good and bad) this drug combination has on you and your HLH.

DETAILED DESCRIPTION:
Hemophagocytic lymphohistiocytosis (HLH) is a rare immunological disorder first recognized almost 70 years ago.(1) Genetic and animal studies have indicated that the familial form of HLH is clearly due to a deficiency of cytotoxic killing. Patients with HLH present with a potentially fatal syndrome of 'hyperimmunity.' These patients have severe inflammation, associated with cytopenias and variably severe bone marrow, liver, or CNS damage. Tissue damage and mortality appear to be due to hypercytokinemia related to persistent immune hyperactivation. An animal model of HLH and correlative human studies all suggest that excessive and abnormal activation of T cells drives the pathophysiology of this disorder, and that suppressing this excessive activation is critical for successful therapy of HLH. It is believed a combination of the two proven induction regimens for hemophagocytic lymphohistiocytosis (HLH) (anti-thymocyte globulin (ATG)- and etoposide-based) will result in response rates and overall survival rates at eight weeks which are comparable or better than the current standard of care (induction therapy per the HLH-94 protocol).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of hemophagocytic lymphohistiocytosis
* Patients <18 years of age
* The patient must have active disease at the time of enrollment
* Patient's legal guardians must sign an Institutional Review Board approved consent form indicating their awareness of the investigational nature and the risks of this study.
* Eligible subjects must be enrolled with the protocol coordinating center

Exclusion Criteria:

* Recent treatment, within 3 months, with another therapeutic regimen for HLH
* Known active malignancy
* Known rheumatologic diagnosis which may be the underlying cause of HLH
* Pregnancy (as determined by serum or urine test) or active breast feeding
* Failure to provide signed informed consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2010-04; Primary Completion 2015-11 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jordan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (15):
- United States (14):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California, San Francisco Department of Pediatrics, San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Nemours, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours, Jacksonville, Florida
  - Florida All Children's Hospital, St. Petersburg, Florida
  - Tulane University Medical Center, New Orleans, Louisiana
  - Children's Hospital Boston, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Cancer Center/Baylor College of Medicine, Houston, Texas
- The Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction Therapy: ATG, rabbit: intravenous, 5 mg/kg/dose, 5 consecutive days Dexamethasone: intravenous, 20mg/m2/day x7days, 10mg/m2/day x7days, 5mg/m2/day x14days, 2.5mg/m2/day x14days, 1.25mg/m2/day x14days Etoposide: intravenous, 150 mg/m2 weekly, starting 7 days after first dose of Thymoglobulin Methotrexate and hydrocortisone: intrathecal to patients with central nervous system involvement, age< 1 yr: 6/8mg (MTX/HC), 1-2 yrs: 8/10mg, 2-3 yrs: 10/12mg, >3 yrs: 12/15 mg, on day 7, 14, 21 and 42
  ATG, rabbit: ATG, rabbit (Thymoglobulin, Genzyme) will be dosed at 5 mg/kg/dose, given IV on 5 consecutive days (titrated over 4 to 8 hours).
  Etoposide: Etoposide will be dosed at 150mg/m2, given IV. The first dose will be given 7 days (+/- 2 days) after the first dose of ATG, and be given weekly for a total of 7 doses.
  Methotrexate: Intrathecal Methotrexate and hydrocortisone will be administered to CNS+ patients.
Period: Treatment Period
Arm/Group | Induction Therapy
Started | 31
Completed | 25
Not Completed | 6
Period: Follow up Until BMT OR 6 Months
Arm/Group | Induction Therapy
Started | 25
Completed | 22
Not Completed | 3
Period: Follow up Until Day 100 Post BMT
Arm/Group | Induction Therapy
Started | 11 (only 11 participants proceeded to BMT; 14 did not)
Completed | 9
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Induction Therapy
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 1
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: To determine the overall survival of patients with hemophagocytic lymphohistiocytosis at 8 weeks after an ATG/etoposide-based induction regimen and to determine the feasibility of this approach in the context of a multicenter clinical trial.
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Therapy
Number analyzed (Participants) | 31
Participants | 25

2. Secondary Outcome: Time to Response
Description: To determine the median time to complete response during 8 weeks of therapy
Time Frame: 8 Weeks
Population: Patients assessed for disease features and classified each week per definition of complete response in order to determine the time at which they achieved complete response.
Measure: Median (Full Range); unit: weeks
Arm/Group | Induction Therapy
Number analyzed (Participants) | 11
weeks | 4 [2 to 7]

3. Secondary Outcome: Overall Survival
Description: To determine overall survival prior to the initiation of BMT (bone marrow transplant) preparative regimen (or day 180, if BMT preparative regimen not yet begun)
Time Frame: up to day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Therapy
Number analyzed (Participants) | 31
Participants | 22

4. Secondary Outcome: Number of Participants Who Experienced Reactivation
Description: To determine the frequency of disease reactivation prior to initiation of BMT preparative regimen (or day 180, if BMT preparative regimen not yet begun)
Time Frame: up to 180 days
Population: all patients surviving to BMT or day 180 and achieving complete or partial response
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Therapy
Number analyzed (Participants) | 21
Participants | 4

5. Secondary Outcome: Overall Survival to Day +100
Description: To determine overall survival to day +100 after BMT, for patients who have undergone BMT within 6 months of study entry
Time Frame: up to day 280
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Therapy
Number analyzed (Participants) | 11
Participants | 9

6. Secondary Outcome: Disease Status at BMT
Description: To determine the rate of complete response at the time of BMT preparative regimen initiation
Time Frame: up to day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Therapy
Number analyzed (Participants) | 11
Participants | 8

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the 8 weeks of the treatment period. All cause mortality was assessed up to day +100 after BMT, if participant proceeded to BMT by day 180. If participant did not proceed to BMT by day 180, all cause mortality was only assessed until day 180.
Arm/Group | Induction Therapy
All-Cause Mortality (participants affected / at risk) | 11/31
Serious Adverse Events (participants affected / at risk) | 22/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Therapy (N=31)
hospitalization (Blood and lymphatic system disorders) | 7 (8)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
acute kidney injury (Renal and urinary disorders) | 3 (3)
status epilepticus (Nervous system disorders) | 1 (1)
multiple organ failure (Vascular disorders) | 4 (4)
herpetic keratitis (Eye disorders) | 1 (1)
hypotension (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Therapy (N=31)
fever (Immune system disorders) | 30 (40)
anemia (Blood and lymphatic system disorders) | 31 (31)
hemorrhage (Blood and lymphatic system disorders) | 5 (5)
hypertension (Vascular disorders) | 3 (3)
thrombosis (Blood and lymphatic system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This is a single arm study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes